CLINICAL TRIAL: NCT00430079
Title: Assessment of Hypoxia in Malignant Gliomas Using EF5
Brief Title: Use of EF5 to Measure the Oxygen Level in Tumor Cells of Patients Undergoing Surgery or Biopsy for Newly Diagnosed Supratentorial Malignant Glioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2012-02419; UPCC# 1301; R21CA093007 (NIH); CDR0000068962 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Diffuse Astrocytoma; Adult Ependymoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Adult Myxopapillary Ependymoma; Adult Oligodendroglioma; Adult Pilocytic Astrocytoma; Adult Pineal Gland Astrocytoma; Adult Subependymoma
MeSH Terms: conditions — Astrocytoma; Ependymoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Glioma, Subependymal | interventions — Etanidazole; Surgical Procedures, Operative; Congresses as Topic

ARMS (1):
- Diagnostic (etanidazole) (Experimental): Patients receive etanidazole derivative EF5 IV over 1-2½ hours once within 1-2 days before surgical resection or biopsy. Tumor tissue, normal tissue, and/or tumor-infiltrated lymph node samples are collected during surgery and stained for biological markers. Fluorescent immunohistochemistry techniques are used to determine the presence, distribution, and levels of EF5 binding.
  Interventions: Drug: etanidazole; Procedure: conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: etanidazole — Given IV
  Other Names: 2-nitro-imidazole derivative; SR-2508
Procedure: conventional surgery — Undergo surgery
  Other Names: surgery, conventional
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial is using EF5 to measure the oxygen level in tumor cells of patients undergoing surgery or surgery biopsy for newly diagnosed supratentorial malignant glioma. Diagnostic procedures using the drug EF5 to measure the oxygen level in tumor cells may help in planning cancer treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the presence and pattern of etanidazole derivative EF5 binding with tumor, based on image and cellular analyses, in patients undergoing surgery or biopsy for newly diagnosed supratentorial malignant gliomas.

II. Determine the level of EF5 binding within histologic subtypes of this tumor in these patients.

Compare the relationship between hypoxia and clinical outcomes in patients with glioblastoma multiforme (GBM) vs non-GBM.

III. Determine the spatial relationships between EF5 binding and tumor tissue biomarkers and pathophysiologic processes (e.g., necrosis, proliferation, and apoptosis) in these patients.

IV. Determine the relationship between EF5 binding and Eppendorf needle electrode measurements in these patients.

OUTLINE:

Patients receive etanidazole derivative EF5 IV over 1-2½ hours once within 1-2 days before surgical resection or biopsy. Tumor tissue, normal tissue, and/or tumor-infiltrated lymph node samples are collected during surgery and stained for biological markers. Fluorescent immunohistochemistry techniques are used to determine the presence, distribution, and levels of EF5 binding.

Patients are followed at 1 month, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study within 1½-2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and/or clinical and imaging evidence of a new brain mass that is likely to be a supratentorial malignant glioma
* Clinical condition and physiologic status indicative of debulking surgery or biopsy as standard initial therapy
* Performance status - Karnofsky performance status 60-100%
* WBC greater than 2,000/mm^3
* Platelet count greater than 90,000/mm^3
* Creatinine less than 2.0 mg/dL
* No significant cardiac condition that would preclude study therapy
* No symptomatic congestive heart failure
* No unstable angina pectoris
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study completion
* Weight no greater than 130 kilograms
* No grade 3 or 4 peripheral neuropathy
* No other invasive malignancy within the past 3 years that is likely to cause a solitary supratentorial metastasis
* No uncontrolled concurrent illness, medical condition, psychiatric illness, or social situation that would preclude study participation
* At least 6 months since prior chemotherapy
* Concurrent corticosteroid therapy allowed
* At least 6 months since prior radiotherapy to lesion or site of lesion
* At least 6 months since prior surgery to lesion or site of lesion except incisional or core biopsy
* Concurrent anticonvulsant therapy allowed
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-07; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Time to local recurrence | Time from study entry (EF5 administration) to local recurrence, assessed up to 3 years

SECONDARY OUTCOMES:
Time to death | Up to 3 years
Presence and pattern of EF5 binding in newly diagnosed brain masses by IHC analyses | At 48 hours after EF5 administration
Levels of EF5 binding within histological subtypes of SMG | At baseline, at 1 hour, and the time of surgery
Relationship between hypoxia and clinical outcomes (i.e., time to local recurrence and survival) | Up to 3 years
  Time to local recurrence and survival will be estimated by the method of Kaplan and Meier.
Association between EF5 binding and Eppendorf needle electrode measurements in brain masses | Up to 3 years
  The correlation between median oxygen pressure (pO2) by Eppendorf electrode measurement and percent of maximal signal in tumors (by EF5 binding) will be assessed by Pearson's correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Judy, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States